CLINICAL TRIAL: NCT00087724
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 2 Study to Evaluate the Safety and Efficacy of FK962 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: A Randomized Study to Evaluate FK962 in Subjects With Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-0-189
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N-(1-acetylpiperidin-4-yl)-4-fluorobenzamide

INTERVENTIONS:
Drug: FK962

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of five fixed dosage levels of FK962 or placebo for 24 weeks in subjects with mild to moderate Alzheimer's disease. Patient visits are every six weeks with limited efficacy measurements at week 6 and 18.

ELIGIBILITY:
Inclusion Criteria:

* Subject satisfies the criteria for the clinical diagnosis of probable AD
* Subject has a score =< 4 on the Modified Hachinski Ischemia Scale at the screening visit

Exclusion Criteria:

* Subject has history or evidence of significant neurologic disease other than AD
* Subject has a history of stroke
* Subject has been treated for schizophrenia or recurrent mood disorder within the previous three years
* Subject has a hematologic or solid malignancy diagnosed within five years prior to study entry
* Subject has medically unstable COPD or asthma
* Subject has end stage CHF (NYHA Class III or IV) or unstable angina
* Subject has evidence of significant renal insufficiency
* Subject has insulin-dependent diabetes mellitus or HbA1C>8.5% at screening

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510
Dates: Start 2004-07; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (81):
- United States (70):
  - Investigational Site, Phoenix, Arizona
  - Sun City, Arizona
  - Investigational Site, Tucson, Arizona
  - Investigational Site, Little Rock, Arkansas
  - Investigational Site, Fresno, California
  - Investigational Site, Irvine, California
  - Investigational Site, Orange, California
  - Investigational Site, San Francisco, California
  - Investigational Site, Sherman Oaks, California
  - Investigational Site, Torrance, California
  - Investigative Site, Denver, Colorado
  - Investigational Site, Denver, Colorado
  - Investigational Site, Darien, Connecticut
  - Investigational Site, Hamden, Connecticut
  - Hamden, Connecticut
  - Investigational Site, Stamford, Connecticut
  - Investigational Site, Fort Myers, Florida
  - Investigational Site, Hialeah, Florida
  - Investigational Site, Hollywood, Florida
  - Investigational Site, Miami, Florida
  - Investigational Site, North Miami, Florida
  - Investigational Site, Ocala, Florida
  - Investigational Site, Port Charlotte, Florida
  - Investigational Site, Sarasota, Florida
  - Investigational Site, Sebring, Florida
  - Investigational Site, Tampa, Florida
  - West Palm Beach, Florida
  - Investigational Site, Snellville, Georgia
  - Snellville, Georgia
  - Investigational Site, Elk Grove, Illinois
  - Investigational Site, Wichita, Kansas
  - Investigational Site, New Orleans, Louisiana
  - Baltimore, Maryland
  - Investigational Site, Newton, Massachusetts
  - Livonia, Michigan
  - Hattiesburg, Mississippi
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Las Vegas, Nevada
  - Investigational Site, Long Branch, New Jersey
  - Investigational Site, Paterson, New Jersey
  - Investigational Site, Piscataway, New Jersey
  - Investigational Site, Albuquerque, New Mexico
  - Investigational Site, Albany, New York
  - Investigational Site, Buffalo, New York
  - Investigational Site, Lawrence, New York
  - Investigational Site, New York, New York
  - Investigational Site, White Plains, New York
  - Charlotte, North Carolina
  - Investigational Site, Centerville, Ohio
  - Investigational Site, Columbus, Ohio
  - Dayton, Ohio
  - Investigational Site, Dayton, Ohio
  - Investigational Site, Toledo, Ohio
  - Investigational Site, Oklahoma City, Oklahoma
  - Investigational Site, Tulsa, Oklahoma
  - Investigational Site, Eugene, Oregon
  - Investigational Site, Medford, Oregon
  - Investigational Site, Bala-Cynwyd, Pennsylvania
  - Investigational Site, Jenkintown, Pennsylvania
  - Investigational Site, Pawtucket, Rhode Island
  - Investigational Site, Johnson City, Tennessee
  - Investigational Site, Nashville, Tennessee
  - Investigational Site, Houston, Texas
  - Investigational Site, San Antonio, Texas
  - Investigational Site, Wichita Falls, Texas
  - Investigational Site, Salt Lake City, Utah
  - Investigational Site, Bennington, Vermont
  - Burlington, Vermont
  - Investigational Site, Norfolk, Virginia
  - Investigational Site, Milwaukee, Wisconsin
- Canada (11):
  - Investigational Site, Kelowna, British Columbia
  - Investigational Site, Penticton, British Columbia
  - Investigational Site, Victoria, British Columbia
  - Investigational Site, Sydney, Nova Scotia
  - Investigational Site, Barrie, Ontario
  - Investigational Site, Greater Sudbury, Ontario
  - Investigational Site, North York, Ontario
  - Investigational Site, Ottawa, Ontario
  - Investigational Site, Toronto, Ontario
  - Investigational Site, Willowdale, Ontario
  - Investigational Site, Regina, Saskatchewan